CLINICAL TRIAL: NCT00581373
Title: Water and the Gastropressor Response - Diurnal Variability (Specific Aim 1.3)
Brief Title: Water and the Gastropressor Response - Diurnal Variability
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Satish R. Raj (Other)
Responsible Party: Sponsor-Investigator, Satish R. Raj, Assistant Professor of Medicine & Pharmacology, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060553; Vanderbilt Discovery (Other: Vanderbilt Univeristy)
Record Dates: First submitted 2007-12-22; First posted 2007-12-27 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Orthostatic Hypotension
Keywords: water; orthostatic hypotension; blood pressure
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): water 16 oz
  Interventions: Other: water 16 fl oz

INTERVENTIONS:
Other: water 16 fl oz — water 16 fl oz in AM and repeat in late afternoon

SUMMARY:
We will test the null hypothesis that there is no diurnal (morning to afternoon)variability in the blood pressure response to the ingestion of water 16 oz.

DETAILED DESCRIPTION:
We will test the null hypothesis that there is no diurnal (morning to afternoon)variability in the blood pressure response to the ingestion of water 16 oz. This will involve having participants ingest 16 oz water rapidly in the morning and in the afternoon.

ELIGIBILITY:
Inclusion Criteria:

* orthostatic intolerance

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-08; Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
blood pressure | 1 day
  peak systolic blood pressure within 60 min of ingestion

SECONDARY OUTCOMES:
heart rate | 1 day
  heart rate at peak BP within 60 min of ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt University Autonomic Dysfunction Center — https://www.vumc.org/autonomic-dysfunction-center/vanderbilt-autonomic-dysfunction